CLINICAL TRIAL: NCT01293240
Title: Prospective Study of Lens Performance of a Monthly Replacement Lens at Two Weeks and Four Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-368-C-400
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-05

CONDITIONS: Myopia; Astigmatism; Presbyopia
MeSH Terms: conditions — Myopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lotrafilcon B (Experimental)
  Interventions: Device: lotrafilcon B contact lens

INTERVENTIONS:
Device: lotrafilcon B contact lens — Commercially marketed, silicone hydrogel contact lens worn bilaterally on a daily wear basis for up to 30 days with a two week and four week evaluation visit.
  Other Names: AIR OPTIX® AQUA, AIR OPTIX® for ASTIGMATISM, AIR OPTIX® AQUA MULTIFOCAL

SUMMARY:
The purpose of this study is to compare the overall performance of a monthly replacement contact lens when worn for one month and when worn for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Habitual and successful wearers of contact lenses made of lotrafilcon B material for at least 4 weeks prior to enrollment.
* Good general health.
* Sphere requirement in the range +6.00 to -10.00 with astigmatism or multifocal correction or no astigmatism or multifocal correction.
* Ability to comply with all protocol-mandated procedures and to attend all scheduled office visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Anterior segment abnormalities (i.e., cataracts, opacities, etc.) or active anterior segment disease.
* Administration of any investigational drug or device within 14 days of study initiation.
* Use of any eye drops with a pharmacological effect within 7 days of Visit 1.
* Known local or systemic hypersensitivity to contact lens cleaning and disinfecting solutions.
* Post-refractive surgery.
* Currently pregnant or lactating by case history.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Lotrafilcon B: Commercially marketed, silicone hydrogel contact lenses worn bilaterally on a daily wear basis for up to 30 days with a two week and four week evaluation visit.
Period: Overall Study
Arm/Group | Lotrafilcon B
Started | 117
Completed | 115
Not Completed | 2
Not completed — Noncompliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 117
Age Continuous [Mean (Standard Deviation); unit: years] — This reporting group includes 114 enrolled and dispensed participants - i.e., 117 total minus 3 missing responses.
  years | 45.8 (12.6)
Gender [Number; unit: participants] — This reporting group includes 115 enrolled and dispensed participants - i.e., 117 total minus 2 missing responses.
  participants
    Female | 79
    Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 2 weeks of wear. Overall comfort was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 2 weeks
Population: Analysis conducted per protocol, with exclusions due to reasons such as protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 8.6 (1.4)

2. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall comfort was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 8.1 (1.7)

3. Primary Outcome: End of Day Dryness
Description: End of day dryness was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 2 weeks of wear. End of day dryness was measured on a 10-point scale, with 1 being very dry and 10 being not dry.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 7.4 (2.1)

4. Primary Outcome: End of Day Dryness
Description: End of day dryness was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. End of day dryness was measured on a 10-point scale, with 1 being very dry and 10 being not dry.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 7.0 (2.4)

5. Primary Outcome: Ocular Redness
Description: Ocular redness was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 2 weeks of wear. Ocular redness was measured on a 10-point scale, with 1 being very red and 10 being not red.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 9.1 (1.4)

6. Primary Outcome: Ocular Redness
Description: Ocular redness was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Ocular redness was measured on a 10-point scale, with 1 being very red and 10 being not red.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 9.0 (1.6)

7. Primary Outcome: Visual Clarity
Description: Visual clarity was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 2 weeks of wear. Visual clarity was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 8.4 (1.5)

8. Primary Outcome: Visual Clarity
Description: Visual clarity was assessed and reported by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Visual clarity was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Units on a scale | 8.2 (1.5)

9. Primary Outcome: Lens Deposits
Description: Protein and lipid deposits on the contact lens surface were assessed for each eye by the investigator using a biomicroscope, which magnifies the appearance of the contact lens on the wearer's eye. Deposits were graded on a scale of 0 to 4, with 0 being none and 4 being severe.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Number analyzed (Eyes) | 223
Units on a scale | 0.6 (0.7)

10. Primary Outcome: Lens Deposits
Description: as for outcome 9
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Number analyzed (eyes) | 224
Units on a scale | 0.8 (0.7)

11. Primary Outcome: Corrected Visual Acuity
Description: Each eye was tested individually while the participant read distant charts in normal lighting. Corrected visual acuity was measured using a Snellen chart, which was converted into logMAR units (logarithm of the minimum angle of resolution). A 20/20 Snellen acuity equates to a logMAR acuity of 0.0 and is considered normal distance eyesight. Positive logMAR values indicate poorer vision, and negative values denote better visual acuity.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Number analyzed (Eyes) | 222
logMAR | 0.04 (0.07)

12. Primary Outcome: Corrected Visual Acuity
Description: as for outcome 11
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Lotrafilcon B
Number analyzed (Participants) | 112
Number analyzed (Eyes) | 223
logMAR | 0.04 (0.08)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial.
Arm/Group | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.